CLINICAL TRIAL: NCT04764175
Title: Assessing Telephone All Nations Breath of Life for Efficacy
Brief Title: Telephone All Nations Breath of Life
Acronym: tANBL
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lehigh University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); University of Kansas Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1612090-2; R01DA048955 (NIH)
Record Dates: First submitted 2021-02-17; First posted 2021-02-21 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Smoking Cessation
Keywords: American Indian; Telephone-Based; Community-Based Participatory Research; Behavioral Intervention
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Intervention Model Description: Bayesian Adaptive Design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telephone All Nations Breath of Life (Experimental): This is a culturally targeted smoking cessation program developed for American Indian communities. It includes individual telephone counseling, text messaging, and educational materials.
  Interventions: Behavioral: Telephone All Nations Breath of Life
- Comparison Program (Active Comparator): This is a non-culturally targeted smoking cessation program. It includes individual counseling, text messaging, and educational materials.
  Interventions: Behavioral: Comparison Program

INTERVENTIONS:
Behavioral: Telephone All Nations Breath of Life — Same as described above.
  Other Names: tANBL
  Arms: Telephone All Nations Breath of Life
Behavioral: Comparison Program — Same as described above.
  Other Names: CP
  Arms: Comparison Program

SUMMARY:
This project formally test an individual, telephone-based version of the All Nations Breath of Life smoking cessation program (tANBL) for American Indians (AI) for efficacy versus an untailored comparison program (CP). The primary outcome is 7-day point prevalence abstinence from smoking cigarettes at 6 months post-baseline. Secondarily, the study examines continuous abstinence and reduction in smoking at both 6 and 12 months post-baseline, as well as demographic predictors of cessation and/or reduction.

DETAILED DESCRIPTION:
The study uses a Bayesian Adaptive Design to examine efficacy of tANBL versus a non-tailored comparison program (CP). All participants will be offered individual telephone counseling, motivational text messaging, educational materials, and the choice of taking pharmacotherapy (must be obtained by participant). Participants in tANBL will receive the culturally tailored versions of all aspects of the program; participants in CP will receive non-tailored versions.

Telephone All Nations Breath of Life (tANBL) Intervention Components

Primary components of tANBL and modifications from the original program are described below:

Individual Sessions: The primary component of tANBL will be a series of individual support sessions, led by an AI facilitator. Community members will be trained in cessation support and counseling. All sessions begin with discussion of individual experiences. All facilitators can be given an extension on the study team's toll-free line, which can be used from any computer. Facilitators will track calls, who participates, how long they last, and recordings (for supervision and training). Facilitators will, in part, use Motivational Interviewing (MI), which has been found effective among AI, enhances motivation for change, and is based on the assumption that many with addictions are not ready to change. The goal is to increase motivation through discrepancy between current behavior and goals/values. The study team developed culturally sensitive counseling scripts to explore positive and negative aspects of, participants' motivation and confidence for quitting smoking, the pros and cons, and plans for change. Participants are asked to identify their values and explore connections between smoking and their ability to live out their values. Participants who score lower on motivation and confidence at each session will be given more Motivational Interviewing.

Text Messaging: Between phone calls, participants receive motivational culturally tailored text messaging, including messages about why smoking is detrimental to health, respecting the sacred nature of tobacco, simple motivational messages to continue trying to quit or stay quit, etc., based on the educational curriculum. The study team has a database of motivational messages developed during the pilot of tANBL; the team will develop and add more messages throughout program implementation to keep messaging relevant and fresh.

Educational Curriculum: The tANBL curriculum includes 11 brochures and combines the latest cessation methods with culturally specific elements, including substantial information about tobacco as a sacred plant for many, though not all, AI tribes, historical trauma, and medical/research mistrust issues, among other topics. Participants have stressed that cultural issues must be ingrained in the program, not given "lip service" with pictures of AI on otherwise "white" materials. Current materials were created by the study team, community advisors, partner organizations, and previous ANBL participants, then sent to an AI graphic artist for layout. Educational materials for this project will be given to participants in paper form based on preferences of pilot participants. Materials are available electronically if a participant wishes.

Pharmacotherapy: Current treatment guidelines suggest pharmacotherapy be offered to all smokers trying to quit; participants have choice of pharmacotherapy, including varenicline, bupropion, nicotine replacement therapy (NRT, patches, gum, or lozenges), a combination, or none, as current best practices suggest. The team considered providing pharmacotherapy as a part of the study, as investigators have done in some previous ANBL studies. However, after discussions with community partners (particularly tribal partners), the team learned that there was a preference for a more real-world scenario where participants can choose to purchase nicotine replacement therapy or see a personal physician for a prescription. Previous ANBL participants have also stated that they would have been able to obtain pharmacotherapy without the study and that provision of it was not a determining factor in taking it. After those discussions, investigators decided to not provide free pharmacotherapy to pilot tANBL participants. Participants were instead given the choice to purchase nicotine replacement therapy or obtain a prescription from personal physicians. Facilitators still discussed all of the available options and allowed participants to ask questions of both facilitators and the study physician to allow for an informed decision. Based on feedback from pilot participants, this was an appropriate approach and will be continued for the efficacy test of tANBL. Investigators will track use of the different types of pharmacotherapy and will examine how it affects quit rates. Facilitators will ask participants who choose not to use any pharmacotherapy about reasons for the choice.

Non-Tailored Comparison Program (CP) Intervention Components

To best test tANBL, we use similar components to the intervention for the CP:

Individual Telephone Sessions: CP arm participants will receive weekly phone calls from non-AI facilitators who will go over similar information using non-tailored materials from the American Cancer Society, through the web portal. Facilitators will not discuss traditional tobacco, historical trauma, or other AI specific topics. They will talk less about social support, as is more common in non-tailored programs.

Text Messaging: CP arm participants will receive non-tailored text messaging.

Educational Curriculum: Non-tailored educational brochures will be provided.

Pharmacotherapy: All participants will be provided with education about pharmacotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Self-reported American Indian
* Smokes at least 1 cigarette per day
* Have a home address or stable address to which we can mail program supplies
* Have a stable telephone number that can be used for the purpose of the study
* Willing to be followed for 12 months

Exclusion Criteria:

* Cannot provide a stable phone number for the purpose of the study that will be available for a minimum of 12 months
* Household member already in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2021-05-13 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Cessation | 6 months
  7-day point prevalence abstinence from smoking cigarettes

SECONDARY OUTCOMES:
Cessation | 12 months
  7-day point prevalence abstinence from smoking cigarettes
Continuous Cessation | 6 months, 12 months
  Continuous abstinence from smoking cigarettes
Smoking Change | 6 months, 12 months
  Change in number of cigarettes per day

CONTACTS AND LOCATIONS:
Overall Officials: Christine M Daley, PhD, MA, SM, Principal Investigator — Lehigh University
Locations (1):
- Lehigh University, Bethlehem, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No